CLINICAL TRIAL: NCT06714565
Title: The Value of Near-infrared Spectroscopy and Blood Pressure Measurements in Estimating Future Fall Risk in Older Adults
Acronym: NIRS-Fall
Status: Recruiting | Type: Observational
Sponsor: Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA) (Other)
Responsible Party: Principal Investigator, Prof. dr. Nathalie van der Velde, Prof., University of Amsterdam
Other Study IDs: NL85457.018.24
Record Dates: First submitted 2024-11-28; First posted 2024-12-03 (Actual); Last update posted 2024-12-19 (Actual); Status verified 2024-12

CONDITIONS: Falls; Orthostatic Hypotension; Older Adults (65 Years and Older)
Keywords: falls; orthostatic hypotension; blood pressure; NIRS; Older adults
MeSH Terms: conditions — Hypotension, Orthostatic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Older adults who have experienced a fall.

SUMMARY:
The investigators aim to study which measurements/definitions from continuous blood pressures measurements (using a Finometer) and from cerebral oxygenation measurements (using near-infrared spectroscopy (NIRS)) are associated with future fall incidents in older adults at risk of falls.

DETAILED DESCRIPTION:
Patients aged 65 years and over with a fall in the last 12 months are eligible for inclusion. After being informed about the study, all participants giving written informed consent will perform the active stand procedure (5min lying, 5 min standing). The hemodynamic measurements that will be performed during this procedure simultaneously consist of:

1. Volume-clamp photoplethysmography on the finger in the digital artery (Finapres medical systems, Enschede, The Netherlands) for continuous blood pressure measurements.
2. PortaLite MKII (Artinis medical systems, Elst, The Netherlands) for continuous cerebral oximetry (NIRS).

After completing the measurements, participants will receive a falls calendar and will be instructed to record falls, fall-related injuries, and fall-related healthcare use on a weekly basis for 12 months.

ELIGIBILITY:
Inclusion Criteria:

* 65 years or older
* History of a fall (in the past year)
* Ability to perform supine-to-stand manoeuvres.
* Ability to sign informed consent.
* a Mini-Mental State Examination (MMSE) score of 21 points or higher or a Montreal Cognitive Assessment (MOCA) - Dutch score of 16 points or higher.
* Sufficient command of the Dutch language

Exclusion Criteria:

* Physically not able to perform sit-to-stand and supine-to-stand manoeuvres.
* Estimated life expectancy of less than one year.

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: Adults aged 65 years and over referred to the outpatient (fall) clinic who have experienced a fall in the past 12 months.
Sampling Method: Non-Probability Sample
Enrollment: 141 (Estimated)
Dates: Start 2024-12-04 (Actual); Primary Completion 2026-12-04 (Estimated); Study Completion 2026-12-05 (Estimated)

PRIMARY OUTCOMES:
Falls during follow-up | From enrollment to 12 months follow-up
  Falls data prospectively collected using fall calenders.

CONTACTS AND LOCATIONS:
Locations (1):
- Amsterdam University Medical Center, location Meibergdreef, Amsterdam, Netherlands

IPD SHARING:
Plan to Share IPD: Undecided